CLINICAL TRIAL: NCT03704337
Title: Effects Of Ingesting A Low Glycemic Whey Protein Energy Bar Prior, During And Following Resistance Exercise And Conditioning On Performance And Recovery
Brief Title: Effects Of Ingesting An Energy Bar On Performance And Recovery
Acronym: NB18
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Richard B. Kreider, Executive Director, Human Clinical Research Facility, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB2017-0602F
Record Dates: First submitted 2018-07-12; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: A randomized, cross-over administration of supplements with approximately 7-10 days between testing sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Commercially Available Food Bar (Experimental): 62 g. Food Bar
  Interventions: Dietary Supplement: Commercially Available Food Bar
- Placebo (Placebo Comparator): 25 g. Dextrose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Commercially Available Food Bar — Active
  Other Names: Food Bar
  Arms: Commercially Available Food Bar
Dietary Supplement: Placebo — Placebo
  Other Names: Dextrose Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of ingesting a low glycemic whey protein energy bar prior, during and following resistance exercise and conditioning on performance and recovery.

DETAILED DESCRIPTION:
Fit-joy is a commercially available food bar marketed as having a low glycemic index and being relatively high in dietary fiber. The fiber contained within this product is isomalto-oligosaccharides (IMO) which is a food ingredient with a relative sweetness level equal to approximately 60% of sucrose. Chemically, IMO is a mixture of glucose oligomers with alpha - (1-6) - linkages. Short and hard exercise produces muscle damage and soreness. The Fit-joy bar contains whey protein that previous research in the investigator's lab showed may be able to decrease the muscle damaging effects of exercise while also helping with muscle growth. The purpose of this study will be to determine if eating a Fit-joy bar before and in the middle of a hard weight training workout will promote positive results during the workout and 48 hours after the workout.

ELIGIBILITY:
Inclusion Criteria:

* Participant is between the ages of 18 and 35
* Participant is apparently healthy
* Participant is involved in a a consistent strength and conditioning program consisting of upper and lower body resistance exercises as well as cardiovascular or sprint conditioning training (for at least the past year for 2-4 days/week), bench press at least your body weight and squat at least 1.5 times your body weight and/or leg press twice your body weight.
* Participant has a Body Mass Index (BMI) < 24.9 or Body Fat Percentage (%BF) < 25.0

Exclusion Criteria:

* Participant has a history of treatment for metabolic disease (i.e., diabetes), hypertension, hypo-tension, thyroid disease, arrhythmia, cardiovascular disease
* Participant has a food allergy (i.e., milk, soy, egg, wheat or nuts)
* Participant uses current prescription medication (birth control is allowed)
* Participant is pregnant or nursing or plans to become pregnant during the next month
* Participant has an intolerance to caffeine and/or other natural stimulants
* Participant has a history of smoking
* Participant drinks excessively (i.e., 12 drinks per week or more)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Glucose Homeostasis: Glucose | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood glucose (mmol/L) obtained from venous blood draws and analyzed General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's).
Glucose Homeostasis: Insulin | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum insulin (µIU/mL) obtained from venous blood draws and analyzed General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's).
Glucose Homeostasis: Insulin to Glucose Ratio | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes the insulin to glucose ratio obtained from venous blood draws and analyzed General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's).
Exercise Glucose Response | Measured at baseline (0-min); 30-min post ingestion of supplement, midway (60-min) and following (90-min) resistance exercise, following sprint condition exercises (110-min), and following post-exercise assessments (130-min) during each treatment.
  Changes in arterialized-venous blood glucose (mmol/L) obtained from a dry finger and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's).

SECONDARY OUTCOMES:
Subjective rating of hypoglycemia | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  A subjective Likert scale that asked participants to rank the frequency and severity of their symptoms of hypoglycemia using the following scale: 0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe). Data will be assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Subjective rating of dizziness | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  A subjective Likert scale that asked participants to rank the frequency and severity of their symptoms of dizziness using the following scale: 0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe). Data will be assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Subjective rating of headaches | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  A subjective Likert scale that asked participants to rank the frequency and severity of their symptoms of headache using the following scale: 0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe). Data will be assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Subjective rating of fatigue | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  A subjective Likert scale that asked participants to rank the frequency and severity of their perceptions of fatigue using the following scale: 0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe). Data will be assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Subjective rating of stomach upset | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  A subjective Likert scale that asked participants to rank the frequency and severity of their symptoms of stomach upset using the following scale: 0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe). Data will be assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Subjective rating of readiness to perform | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  A subjective Likert scale assessing readiness to perform on a visual analog scale (VAS) measured prior to supplementation, following exercise, and after 48 hours of recovery from exercise. The scale ranges from "1" - strongly disagree they are ready to perform to "5" - they strongly agree they are ready to perform. Data will be assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Subjective rating of pain | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  A subjective Likert scale that assessed perceptions of pain in response the application of a standard amount of pressure applied using an algometer and measured prior to supplementation, following exercise, and after 48 hours of recovery from exercise. The scale was a straight horizontal-line with no hash-markings only wording beneath the line, which read from left-to-right "no pain, dull ache, slight pain, more slight pain, painful, very painful, and unbearable pain". Participants were instructed to scribe one clear mark bisecting the line which represented their pain level the best for each of the three pressure application sites. A ruler was used to measure the participant's mark from the left-to-right in cm and was recorded in the data as such numerical value. Data will be assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Agility Performance Time | Measured 30-min after ingestion of supplement and after performing 60-min of resistance exercise during each treatment.
  Time in seconds to perform 3 sprints around 4 cones for the Nebraska Agility Drill (NAD) with 30-seconds recovery. The tests were performed after completing the resistance exercise once during each treatment. Individual and cumulative performance times were assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Sprint Performance Times | Measured 30-min after ingestion of supplement and after performing 60-min of resistance exercise during each treatment.
  Measured as the time (in seconds) it takes to sprint three 40-yard dashes with 30-seconds recovery. The tests were performed after completing the resistance exercise once during each treatment. Individual and cumulative performance times will be assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Maximal voluntary muscle contraction (MVC) leg extension torque | Measured prior to supplementation, following 30-min rest and 80-min of exercise, and after 48 hours of recovery from exercise during each treatment.
  Measured using a Kin-Com isokinetic dynamometer and expressed in Newton meters assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Maximal voluntary muscle contraction (MVC) leg extension force | Measured prior to supplementation, following 30-min rest and 80-min of exercise, and after 48 hours of recovery from exercise during each treatment.
  Measured using a Kin-Com isokinetic dynamometer and expressed in Newtons assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Maximal voluntary muscle contraction (MVC) leg extension power | Measured prior to supplementation, following 30-min rest and 80-min of exercise, and after 48 hours of recovery from exercise during each treatment.
  Measured using a Kin-Com isokinetic dynamometer and expressed in Watts assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Maximal voluntary muscle contraction (MVC) leg extension work | Measured prior to supplementation, following 30-min rest and 80-min of exercise, and after 48 hours of recovery from exercise during each treatment.
  Measured using a Kin-Com isokinetic dynamometer and expressed in Joules assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Maximal voluntary muscle contraction (MVC) leg flexion torque | Measured prior to supplementation, following 30-min rest and 80-min of exercise, and after 48 hours of recovery from exercise during each treatment.
  Measured using a Kin-Com isokinetic dynamometer and expressed in Newton Meters assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Maximal voluntary muscle contraction (MVC) leg flexion force | Measured prior to supplementation, following 30-min rest and 80-min of exercise, and after 48 hours of recovery from exercise during each treatment.
  Measured using a Kin-Com isokinetic dynamometer and expressed in Newtons assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Maximal voluntary muscle contraction (MVC) leg flexion power | Measured prior to supplementation, following 30-min rest and 80-min of exercise, and after 48 hours of recovery from exercise during each treatment.
  Measured using a Kin-Com isokinetic dynamometer and expressed in Watts assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Maximal voluntary muscle contraction (MVC) leg flexion work | Measured prior to supplementation, following 30-min rest and 80-min of exercise, and after 48 hours of recovery from exercise during each treatment.
  Measured using a Kin-Com isokinetic dynamometer and expressed in Joules assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Markers of Catabolism: Blood Urea Nitrogen | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood urea nitrogen in mmol/L (BUN) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Markers of Catabolism: Creatinine | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood creatinine (umol/L) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Markers of Catabolism: Lactate Dehydrogenase | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood LDH (IUl/L) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Markers of Catabolism: Creatine Kinase | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood CK (IUl/L) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Markers of Catabolism: BUN/Creatinine Ratio | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood BUN/creatinine ratio obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Stress and Sex Hormones: Cortisol | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood cortisol (ug/dL) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Stress and Sex Hormones: Testosterone | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood testosterone (ng/mL) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Stress and Sex Hormones: Cortisol to Testosterone Ratio | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in the ratio of cortisol to testosterone obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Markers of Inflammation: Interferon Gama (IFNy) | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood IFNy (pg/mL) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Markers of Inflammation: Interleukin-13 (IL-13) | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood IL-13 (pg/mL) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Markers of Inflammation: Interleukin-1 beta (IL-1ß) | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood IL-1ß (pg/mL) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Markers of Inflammation: Interleukin-4 beta (IL-4) | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood IL-4 (pg/mL) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Markers of Inflammation: Interleukin-6 beta (IL-6) | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood IL-6 (pg/mL) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Markers of Inflammation: Interleukin-8 beta (IL-8) | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood IL-8 (pg/mL) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).
Markers of Inflammation: Tumor Necrosis Factor alpha (TNFα) | Measured prior to supplementation (Pre), 30-min after ingestion of supplement and after performing the 80-min exercise bout (Post-Exercise), and after 48 hours of recovery from exercise bout (Recovery) during each treatment.
  Changes in serum blood TNFα (pg/mL) obtained from venous blood draws and assessed via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's).

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Exercise & Sport Nutrition Lab - Human Clinical Research Facility, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grubic TJ, Sowinski RJ, Nevares BE, Jenkins VM, Williamson SL, Reyes AG, Rasmussen C, Greenwood M, Murano PS, Earnest CP, Kreider RB. Comparison of ingesting a food bar containing whey protein and isomalto-oligosaccharides to carbohydrate on performance and recovery from an acute bout of resistance-exercise and sprint conditioning: an open label, randomized, counterbalanced, crossover pilot study. J Int Soc Sports Nutr. 2019 Aug 13;16(1):34. doi: 10.1186/s12970-019-0301-z. PMID 31409363